CLINICAL TRIAL: NCT00271570
Title: Infliximab (Remicade) for Patients With Acute Kawasaki Disease Who Fail to Become Afebrile After Intravenous Gamma Globulin Therapy
Brief Title: Infliximab (Remicade) for Patients With Acute Kawasaki Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Jane C. Burns, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 041374; 2004-0548
Record Dates: First submitted 2005-12-30; First posted 2006-01-02 (Estimated); Results first posted 2009-12-29 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2009-11

CONDITIONS: Kawasaki Disease
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Infliximab; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Second Dose of IVIG (2g/kg) (Active Comparator): Subjects who did not respond to the first dose of IVIG received a 2nd dose of IVIG in this arm (2g/kg)
  Interventions: Biological: Intravenous immunoglobulin (IVIG)
- Infliximab (5mg/kg) (Experimental): Remicade (5mg/kg) single dose
  Interventions: Drug: Infliximab (Remicade)

INTERVENTIONS:
Drug: Infliximab (Remicade) — Remicade was 5 mg/kg IV (single dose)
  Arms: Infliximab (5mg/kg)
Biological: Intravenous immunoglobulin (IVIG) — 2nd dose of IVIG (2g/kg)
  Other Names: Gammagard, Gamunex
  Arms: Second Dose of IVIG (2g/kg)

SUMMARY:
This study evaluates the safety of infliximab in infants and children with acute Kawasaki Disease.

DETAILED DESCRIPTION:
This study is an exploratory, pilot study to examine tolerance and pharmacokinetics of infliximab in infants and children with acute Kawasaki Disease.

ELIGIBILITY:
Inclusion criteria

To be eligible for the trial, subjects must meet all of the following criteria:

1. All eligible subjects, or legal representative, must provide written informed consent/assent, prior to initiation of any study procedure.
2. Eligible subjects will be infants and children, under 18 years old, with acute KD who remain or become febrile (>/= 38.3˚ C or 101.0˚ F) after the end of the 48 h-period after completing their IVIG infusion (2gm/kg).
3. Patients must have persistent or reoccurrence of fever > 48 hours of observation to be eligible for the trial.
4. Prior to the initial IVIG treatment, patients must have been febrile for >/= 3 days and have met 4/5 standard clinical criteria (Table 1) - OR - patients with fever and 3/5 clinical criteria will be eligible if echocardiogram demonstrates at least one coronary artery segment with a Z score of > 2.
5. Patients must present for their initial diagnosis and IVIG treatment within the first 14 days after fever onset (Illness Day 14).
6. Females of childbearing potential and males must be using adequate contraception (abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, or surgical sterilization) throughout the trial.
7. All eligible subjects must have a chest radiograph within one week prior to first infusion of study drug with no evidence of malignancy, infection or fibrosis.

Exclusion criteria

If a subject has any of the following criteria, he or she may not be enrolled in the study:

1. Have been receiving corticosteroids (ie, via any route) at doses > 1 mg/kg prednisone equivalent daily.
2. Have history of TB or TB exposure.
3. Have history of histoplasmosis or coccidiomycosis.
4. Have received anakinra (Kineret®), etanercept (Enbrel®), or adalimumab (Humira®) within 1 month prior to first study drug administration.
5. Have any chronic disease, except asthma, atopic dermatitis or controlled seizure disorder.
6. Have documented history of current active hepatitis B or a history of hepatitis C infection.
7. Have documented history of human immunodeficiency virus (HIV) infection
8. Have received a transplanted organ (with the exception of a corneal transplant performed > 3 months prior to first study drug administration).
9. Have a known malignancy or history of malignancy within the 5-year period prior to first study drug administration (with the exception of squamous or basal cell carcinoma of the skin that has been completely excised without evidence of recurrence).
10. Have a history of prior lymphoproliferative disease including lymphoma.
11. Have multiple sclerosis or other central demyelinating disorder.
12. Have received any previous treatment with infliximab or other monoclonal antibodies.
13. Have used any investigational drug within 1 month prior to first study drug administration or within 5 half-lives of the investigational agent, whichever is longer.
14. Are participating in another investigative trial, involving investigational agents, during participation in this trial.
15. Have a history of substance abuse (drug or alcohol) within the previous 3 years.
16. Are pregnant, nursing, or planning pregnancy (both men and women) during the trial or within the 6-month period thereafter.
17. Have a known allergy to murine proteins or other chimeric proteins.
18. Patients with ischemic congestive heart failure.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2004-04; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane C Burns, M.D., Principal Investigator — UCSD/CHHC
Locations (1):
- Ucsd/Chhc, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- IVIG Arm (2 gr/kg): 2nd dose of IVIG (2gr/kg)
- Infliximab (5mg/kg): Remicade (Infliximab Arm of 5mg/kg)
Period: Overall Study
Arm/Group | IVIG Arm (2 gr/kg) | Infliximab (5mg/kg)
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IVIG Arm (2 gr/kg) | Infliximab (5mg/kg) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 12 | 24
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 1.833 (.3) | 1.667 (.3) | 1.75 (.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events (Focused on Side Effects From IVIG or Infliximab Administration)
Description: The safety of giving infliximab to treat IVIG-resistant Kawasaki disease was measured by recording the number of adverse events that occurred in each group. An adverse event (AE) was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of either IVIG or infliximab, regardless of whether it was considered related to IVIG or infliximab, that occured during the course of this study.In particular we evaluated for AEs related to side effects from infliximab or IVIG.
Time Frame: 2 weeks
Measure: Number; unit: events
Arm/Group | IVIG Arm (2 gr/kg) | Infliximab (5mg/kg)
Number analyzed (Participants) | 12 | 12
events | 2 | 3

2. Primary Outcome: Area Under the Curve of Infliximab Concentration Before Infliximab Infusion and Then 2 and 24 Hours, 1 Week (5 to 9 Days), 2 Weeks (12 to 16 Days), and 4 Weeks (26 to 30 Days) After Infliximab Infusion)
Description: The area under the curve (AUC) from time 0 to the last measurable concentration (AUC0-last) was estimated using the trapezoidal rule up to the last measurable concentration.Samples were collected before infliximab infusion and then at 2 and 24 hours, 1 week (5 to 9 days), 2 weeks (12 to 16 days), and 4 weeks (26 to 30 days) after infliximab infusion. Subjects with detectable infliximab concentrations at week 4 had another sample drawn at week 10 (68 to 72 days).
Time Frame: before infliximab infusion and then 2 and 24 hours, 1 week (5 to 9 days), 2 weeks (12 to 16 days), and 4 weeks (26 to 30 days) after infliximab infusion.
Measure: Median (Inter-Quartile Range); unit: micogram*day/ml
Arm/Group | IVIG Arm (2 gr/kg) | Infliximab (5mg/kg)
Number analyzed (Participants) | 12 | 12
micogram*day/ml | 0 [0 to 0] | 619 [458 to 891]

ADVERSE EVENTS:
Arm/Group | IVIG Arm (2 gr/kg) | Infliximab (5mg/kg)
Serious Adverse Events (participants affected / at risk) | 2/12 | 3/12
Other Adverse Events (participants affected / at risk) | 8/12 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVIG Arm (2 gr/kg) (N=12) | Infliximab (5mg/kg) (N=12)
Cerebellar ataxia (Nervous system disorders) | 0 (0) | 1 (1) — Acute cerebellar ataxia attributed to KD (resolved); giant aneurysms (> 8 mm) treated with warfarin (z-max: RCA, 15.8; LAD, 7.44)
Enlarging aneurysms (Cardiac disorders) | 0 (0) | 1 (1) — Enlarging aneurysms (z-max: RCA, 7.5; LAD, 4.9); readmitted for repeat infliximab and IVIG infusion; aneurysms resolved
Fever (General disorders) | 1 (1) | 0 (0) — Persistent fever plus rising CRP treated with IV methylprednisilone; aneurysms of RCA and LAD (z-max: RCA, 7.2; LAD, 8.1)
Persistent Fever (General disorders) | 1 (1) | 0 (0) — Persistent fever treated with IV methylprednisilone, oral steroids, and methotrexate; dilated coronary arteries (z-max: RCA, 4.6; LAD, 3.3), dilatation resolved
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Drug-related rash with eosinophilia and systemic symptoms, attributed to azithromycin administered before study entry (reported to the FDA), requiring hospitalization for supportive care; normal coronary arteries
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVIG Arm (2 gr/kg) (N=12) | Infliximab (5mg/kg) (N=12)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute gastroentiritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Secondary to rotavirus
Allergic rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Ankle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bee sting (General disorders) | 1 (1) | 0 (0)
Conjunctival injection (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Coronary artery aneurysm (Cardiac disorders) | 1 (1) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heart murmur (Cardiac disorders) | 1 (1) | 1 (1) — I/VI systolic ejection murmur
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 3 (3) | 3 (3)
High pitched crying (General disorders) | 0 (0) | 1 (1) — Sometimes raspy voice
Hoarseness (General disorders) | 0 (0) | 1 (1)
IV infiltrate (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Interval increase in size of coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Irregular heart rate (Cardiac disorders) | 1 (1) | 0 (0)
Lip laceration from accidental trauma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Lung infiltrate (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pain (Nervous system disorders) | 1 (1) | 1 (1)
Peeling of fingers and toes (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Peeling of hands (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) — Trivial size
Phimosis with swelling of foreskin (Renal and urinary disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Steven's Johnson Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Teary eyes (Eye disorders) | 1 (1) | 0 (0)
Temperature of 99.5 F (General disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No